CLINICAL TRIAL: NCT02662023
Title: Continuous Transversus Abdominis Plane Nerve Blocks: Relative Effects of a Basal Infusion vs. Repeated Bolus Doses (A Randomized, Double-Masked, Active-Control, Split-Body, Crossover Study)
Brief Title: Continuous TAP Blocks: Relative Effects of a Basal Infusion vs. Repeated Bolus Doses
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Zyno Medical (Industry); Teleflex (Industry)
Responsible Party: Principal Investigator, Brian M. Ilfeld, MD, MS, Professor of Anesthesiology, In Residence, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TAP Basal vs. Bolus
Record Dates: First submitted 2016-01-20; First posted 2016-01-25 (Estimated); Results first posted 2021-03-18 (Actual); Last update posted 2021-03-18 (Actual); Status verified 2021-02

CONDITIONS: Postoperative Pain
Keywords: Healthy Human Volunteers
MeSH Terms: conditions — Pain, Postoperative | interventions — NOP-bolus regimen

STUDY DESIGN:
Intervention Model Description: This is a split-body study in which each study subject receives both treatments: one on each side of the body. Which treatment is applied to which side of the body is randomized (and masked).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The only individual aware of the treatment group assignments is the investigational pharmacist who has no interaction with the study subjects. Treatment group assignments were released by the investigational pharmacy only after completion of data collection.
Oversight: Data Monitoring Committee: No

ARMS (2):
- RIGHT side BOLUS and left side basal (Experimental): Bilateral transversus abdominis catheters were inserted and ropivacaine 0.2% administered concurrently. For the right catheter, the ropivacaine was administered as two separate bolus doses of 24 mL each: one at time point zero and one 3 hours later. For the left catheter, the ropivacaine was administered as a continuous basal infusion (8 mL/h) from time point zero for the following 6 hours
  Interventions: Drug: Bolus; Drug: Basal
- RIGHT side BASAL and left side bolus (Active Comparator): Bilateral transversus abdominis catheters were inserted and ropivacaine 0.2% administered concurrently. For the right catheter, the ropivacaine was administered as a continuous basal infusion (8 mL/h) from time point zero for the following 6 hours. For the left catheter, the ropivacaine was administered as two separate bolus doses of 24 mL each: one at time point zero and one 3 hours later
  Interventions: Drug: Bolus; Drug: Basal

INTERVENTIONS:
Drug: Bolus — A transversus abdominis catheter was inserted and ropivacaine 0.2% administered as two separate bolus doses of 24 mL each: one at time point zero and one 3 hours later.
  Other Names: automatic intermittent bolus doses
Drug: Basal — A transversus abdominis catheter was inserted and ropivacaine 0.2% administered as a continuous basal infusion (8 mL/h) from time point zero for the following 6 hours.
  Other Names: continuous basal infusion

SUMMARY:
Single-injection transversus abdominis plane (TAP) blocks have been used to treat postoperative pain, and are become very popular within the United States because of their high analgesic potency and relative ease of placement. Unfortunately, the longest local anesthetic available lasts only 8-12 hours. Continuous TAP blocks-also termed "perineural infusion"-involve bathing the multiple nerves of the abdominal wall in local anesthetic using a percutaneously-inserted perineural catheter inserted just anterior (ventral) and cephalad to the anterior superior iliac spine. For most catheter locations, an infusion is preferred to a single-injection nerve block because the duration of analgesia may be extended to better match the duration of surgical pain. But, unlike brachial plexus, femoral, and sciatic nerve perineural infusion, a continuous basal infusion of local anesthetic does not provide adequate analgesia for TAP catheters. This may be due to the fact that the TAP is a relatively tight space, so it might require a bolus of fluid to adequately spread the perineural local anesthetic to the multiple required nerves (as evidence of this, single-injection TAP blocks are very effective, although with a limited duration). The result is that while single-injection TAP blocks are widely used, TAP catheters have not been adopted. This scenario leaves surgical pain untreated following the resolution of the single-injection TAP block. The recent development of an infusion pump that can automatically deliver repeated bolus doses may allow the spread of local anesthetic to the multiple sensory nerves necessary to provide adequate analgesia, with a duration that better matches postoperative requirements. The investigators therefore propose a randomized, double-masked, controlled trial to determine if delivering local anesthetic as a repeated bolus dose results in improved local anesthetic spread/effects compared with a continuous basal infusion for TAP catheters.

DETAILED DESCRIPTION:
This investigation will be a randomized, observer-masked, controlled, split-body, human-subjects clinical trial. Of note, the investigators will be using standard-of-care local anesthetics under their FDA approved purpose and do not plan to research a possible change of indication or use of these drugs as part of this research project.

Volunteers will be solicited using the CTRI Research Match and an existing database of volunteers (IRB approved). If a volunteer meets inclusion/exclusion criteria (see Eligibility Criteria) and desires study participation, written, informed consent will be obtained using a UCSD IRB-approved/stamped ICF. A urine pregnancy test will be administered to all women of childbearing age following written informed consent but before any study interventions. This urine test will be administered by CTRI nursing staff using standard, FDA-approved urine pregnancy testing devices.

Perineural catheter insertion: Following written, informed consent, subjects will be admitted to the UCSD CTRI Center for Clinical Research Services (CCR) and have demographic/morphometric data recorded (e.g., age, weight, height). An intravenous line will be placed in an upper extremity, followed by external monitors (pulse oximeter, blood pressure, and EKG), and oxygen by nasal cannula. Sedation will be provided with intravenous fentanyl (50 μg) and/or midazolam (1 mg). Bilateral TAP perineural catheters (FlexBlock, Teleflex Medical, Reading, PA, USA) will be inserted using ultrasound guidance using a technique previously described. To check the perineural catheter placement accuracy, 5 mL of normal saline will be administered via the catheters under ultrasound guidance with the definition of a successful catheter insertion an increase in fluid volume within the TAP (the plane between the transversus abdominis muscle and internal oblique muscle). Inaccurately inserted catheters will be replaced.

Treatment Group Assignment: Subjects will act as their own controls: the right side will be randomized to one of two treatment groups: ropivacaine 0.2% administration as either a basal infusion (8 mL/h) or bolus doses (24 mL administered every 3 hours). The left side will receive the other possible treatment. Randomization will be based on computer-generated codes. Randomization will be in blocks of four. An infusion pump with study infusate will be attached to each of the perineural catheters and initiated at Hour 0. Which side of the participant's body will receive the basal rate and which side will receive bolus volume will depend upon the treatment group assignment but the total dose of local anesthetic is the same for each side.

The tubing from the pumps to the subjects will be gently wound at least 5 rotations and covered with opaque tape, masking which perineural catheter is receiving which treatment (ropivacaine is clear, so the flow through the clear tubing from the tape to the perineural catheters will not be visually distinguishable).

Local Anesthetic Administration: The infusion pump administering the basal infusion will be initiated at Hour 0. The infusion pump administering bolus doses will administer a 24 mL bolus dose every 3 hours beginning at Hour 0. Perineural catheters will be removed after 6 hours (a total of 2 bolus doses).

Food and Drink: Both food and accompanying beverages/water will be provided by the hospital and served by the nursing staff immediately following catheter insertion. Meals will be provided without charge to the study subjects. There is no restriction on oral intake following catheter insertion. Subjects will remain within the CTRI-CCR until catheter withdrawal.

Outcome measurements: At all time points, the right side will be measured first, followed by the left side (subjects in the supine position).

Measurements will be performed at baseline (prior to local anesthetic administration), after 6 hours of administration, and at each hour in between for a total of 7 time points:

* Hour 0 (baseline) just prior to local anesthetic administration
* Hours 1 and 2
* Hour 3, just prior to the scheduled bolus dose at Hour 3
* Hours 4 and 5
* Hour 6

The sensory deficit will be measured using two methods:

* von Frey filaments (mechanical detection threshold)
* Cold roller (cold deficit)

The sensory deficit will be measured along two separate anatomical lines at each time point:

* The mid-axillary "vertical" line (measuring cephalad-caudad effects)
* A transverse "horizontal" line passing through the anterior superior iliac spine (measuring anterior-posterior effects)

Statistical analysis: The investigators' calculations are focused on the primary hypothesis that when using transversus abdominis plane (TAP) block perineural catheters, providing local anesthetic in repeated bolus doses increases the cephalad-caudad local anesthetic effects compared with a basal-only infusion of the same volume and dose of local anesthetic. To measure cephalad-caudad local anesthetic effects, we will measure the cephalad-caudad sensory deficit to cold temperature in centimeters along the mid-axillary line. The primary end point will be this measurement after 6 hours of local anesthetic administration (6 hours of a continuous basal infusion or 2 bolus doses at 3-hour increments, the last being 3 hours prior to the measurement of the primary endpoint). Each subject will act as their own control with each side receiving a different treatment. Normality of distribution will be determined using the Shapiro-Wilk normality test (Prism 6, GraphPad, San Diego, California). For normally distributed data, comparisons for parametric and nonparametric data will be tested using the t-test or Mann-Whitney test and presented as mean (SD) or median [interquartile], respectively. Nominal data will be analyzed using the Pearson Chi square test. P<0.05 will be considered significant.

Sample size estimation: With 21 evaluable subjects we will have 80% power at the 0.05 significance level to detect the superiority of the administration of local anesthetic as repeated bolus doses as compared with a continuous basal infusion at Hour 6 (primary outcome). Using an expected standard deviation of 7 cm for the primary endpoint, and given a 2-sided Type I error protection of 0.05 and power=0.80, approximately 21 subjects in each treatment arm will be required to detect a difference between treatment group means of 6 cm. Since this is a split-body study design and each subject will have one of each treatments on opposite sides of the body, 21 subjects total will produce 21 subjects in each treatment arm. The investigators chose 6 cm as a detectable treatment difference because a 3 cm distance is approximately equivalent to the width of one dermatome, and the vast majority of anesthesiologists would consider a 2-dermatome difference clinically significant. To allow for a larger-than-anticipated standard deviations, smaller-than-anticipated difference between treatment means, drop out subjects, or failed catheters, the investigators will enroll a total of 24 subjects.

ELIGIBILITY:
Inclusion Criteria:

1. healthy volunteers weighing more than 45 kg;
2. must be willing to have bilateral transverses abdominis plane nerve block catheters be placed with subsequent ropivacaine administration and sensory testing for 6 hours

Exclusion Criteria:

1. BMI greater than 40 (BMI=weight in kg/ [height in meters];
2. regular opioid use within the previous 2 months;
3. previous participation within the same study;
4. allergy to study medications;
5. known renal insufficiency (creatinine > 1.5 mg/dL);
6. pregnancy;
7. incarceration; and
8. any known neuro-muscular deficit of either abdominal wall.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2016-02; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian Ilfeld, MD, MS, Principal Investigator — University of California, San Diego
Locations (1):
- Ucsd Ctri, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ilfeld BM. Continuous peripheral nerve blocks: a review of the published evidence. Anesth Analg. 2011 Oct;113(4):904-25. doi: 10.1213/ANE.0b013e3182285e01. Epub 2011 Aug 4. PMID 21821511
- [Background] Hebbard PD, Barrington MJ, Vasey C. Ultrasound-guided continuous oblique subcostal transversus abdominis plane blockade: description of anatomy and clinical technique. Reg Anesth Pain Med. 2010 Sep-Oct;35(5):436-41. doi: 10.1097/aap.0b013e3181e66702. PMID 20830871
- [Background] Stoving K, Rothe C, Rosenstock CV, Aasvang EK, Lundstrom LH, Lange KH. Cutaneous Sensory Block Area, Muscle-Relaxing Effect, and Block Duration of the Transversus Abdominis Plane Block: A Randomized, Blinded, and Placebo-Controlled Study in Healthy Volunteers. Reg Anesth Pain Med. 2015 Jul-Aug;40(4):355-62. doi: 10.1097/AAP.0000000000000252. PMID 25923818
- [Background] Borglum J, Jensen K, Christensen AF, Hoegberg LC, Johansen SS, Lonnqvist PA, Jansen T. Distribution patterns, dermatomal anesthesia, and ropivacaine serum concentrations after bilateral dual transversus abdominis plane block. Reg Anesth Pain Med. 2012 May-Jun;37(3):294-301. doi: 10.1097/AAP.0b013e31824c20a9. PMID 22476239
- [Background] Carney J, Finnerty O, Rauf J, Bergin D, Laffey JG, Mc Donnell JG. Studies on the spread of local anaesthetic solution in transversus abdominis plane blocks. Anaesthesia. 2011 Nov;66(11):1023-30. doi: 10.1111/j.1365-2044.2011.06855.x. Epub 2011 Aug 18. PMID 21851346
- [Result] Khatibi B, Said ET, Sztain JF, Monahan AM, Gabriel RA, Furnish TJ, Tran JT, Donohue MC, Ilfeld BM. Continuous Transversus Abdominis Plane Nerve Blocks: Does Varying Local Anesthetic Delivery Method-Automatic Repeated Bolus Versus Continuous Basal Infusion-Influence the Extent of Sensation to Cold?: A Randomized, Triple-Masked, Crossover Study in Volunteers. Anesth Analg. 2017 Apr;124(4):1298-1303. doi: 10.1213/ANE.0000000000001939. PMID 28319550

RESULTS

PARTICIPANT FLOW:
Groups:
- Right Side of the Body Randomized to Bolus: Ropivacaine 0.2% administration as repeated, scheduled (one/3 h) bolus doses (24 mL) x 6 h
  Perineural ropivacaine administration.
  Since it's a split body study ,left side of the body of these participants received Ropivacaine 0.2% perineural administration as a continuous basal infusion (8 mL/h) x 6 h.
- Right Side of the Body Randomized to Basal: Ropivacaine 0.2% administration as a continuous basal infusion (8 mL/h) x 6 h
  Perineural ropivacaine administration.
  Since it's a split body study, left side of these participants received Ropivacaine 0.2% administration as repeated, scheduled (one/3 h) bolus doses (24 mL) x 6 h
Period: Overall Study
Arm/Group | Right Side of the Body Randomized to Bolus | Right Side of the Body Randomized to Basal
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Since it's a split body study, right side of each participant's body was randomized to bolus or basal arm. Left side of same participant's body simultaneously received the opposite treatment of what the right side of the body was randomized to( for example: if right side of one participants body was randomized to Bolus doses then the left side of the same participant's body received ropivacaine administration as basal infusion).
Groups:
- Right Side of the Body Randomized to Bolus: Ropivacaine 0.2% administration as repeated, scheduled (one/3 h) bolus doses (24 mL) x 6 h
  Perineural ropivacaine administration.
  Since it's a split body study ,left side of the body of these participants simultaneously received Ropivacaine 0.2% perineural administration as a continuous basal infusion (8 mL/h) x 6 h.
- Right Side of the Body Randomized to Basal: Ropivacaine 0.2% administration as a continuous basal infusion (8 mL/h) x 6 h
  Perineural ropivacaine administration.
  Since it's a split body study, left side of these participants simultenously received Ropivacaine 0.2% administration as repeated, scheduled (one/3 h) bolus doses (24 mL) x 6 h.
- Total: Total of all reporting groups
Arm/Group | Right Side of the Body Randomized to Bolus | Right Side of the Body Randomized to Basal | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 12 | 24
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.2 (14.0) | 36.6 (9.6) | 35 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 7 | 7 | 14
Region of Enrollment [Number; unit: participants]
  United States | 12 | 12 | 24
Height [Mean (Standard Deviation); unit: cm] | 167.9 (8.9) | 175.7 (6.5) | 172 (9)
Weight [Mean (Standard Deviation); unit: kg] | 80.0 (26.4) | 74.9 (11.7) | 77 (20)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 28.3 (8.9) | 24.3 (3.6) | 26 (7)

OUTCOME MEASURES:

1. Primary Outcome: Sensory Deficit (Cold Roller), Mid-axillary Line
Description: The distance of sensory deficit to cold measured in centimeters along the mid-axillary line. A cold roller is a device that looks like a paint application roller, but the roller itself is metal that can be brought to freezing. It is placed in the mid-axillary line and moved up and down until the sensory deficit to cold is revealed and subsequently measured.
Time Frame: 6 hours following the initiation of local anesthetic administration
Measure: Mean (Standard Deviation); unit: cm
Groups:
- Bolus: ropivacaine 0.2% administration as repeated, scheduled (one/3 h) bolus doses (24 mL) x 6 h
  perineural ropivacaine administration
- Basal: ropivacaine 0.2% administration as a continuous basal infusion (8 mL/h) x 6 h
  perineural ropivacaine administration
Arm/Group | Bolus | Basal
Number analyzed (Participants) | 24 | 24
cm | 9.2 (5.6) | 9.3 (5.1)

2. Secondary Outcome: Sensory Deficit (Cold Roller), Mid-axillary Line
Description: as for outcome 1
Time Frame: Hourly from Hours 0-5 following the initiation of local anesthetic administration
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Bolus | Basal
Number analyzed (Participants) | 24 | 24
cm
  Hour 0 | 0 (0.3) | 0 (0)
  Hour 1 | 8.0 (5.7) | 2.9 (4.2)
  Hour 2 | 8.6 (5.2) | 7.8 (6.4)
  Hour 3 | 7.8 (6.2) | 7.5 (4.2)
  Hour 4 | 9.3 (5.7) | 9.0 (6.2)
  Hour 5 | 9.3 (5.9) | 9.7 (4.9)

3. Secondary Outcome: Sensory Deficit (Cold Roller), Transverse Horizontal Line
Description: The distance of sensory deficit to cold measured in centimeters along the transverse horizontal line passing through the anterior superior iliac spine. A cold roller is a device that looks like a paint application roller, but the roller itself is metal that can be brought to freezing. It is placed along the line described above and moved anterior and posterior until the sensory deficit to cold is revealed and subsequently measured.
Time Frame: Hourly from Hours 0-6 following the initiation of local anesthetic administration
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Bolus | Basal
Number analyzed (Participants) | 24 | 24
cm
  Hour 0 | 0 (0) | 0 (0)
  Hour 1 | 11.8 (7.6) | 7.7 (10.5)
  Hour 2 | 14.0 (7.9) | 14.3 (11.5)
  Hour 3 | 15.6 (10.8) | 14.4 (9.0)
  Hour 4 | 16.1 (8.9) | 15.4 (8.3)
  Hour 5 | 16.6 (9.3) | 15.3 (9.3)
  Hour 6 | 16.8 (9.6) | 15.8 (8.1)

4. Secondary Outcome: Sensory Deficit (Von Frey Hairs), Transverse Horizontal Line
Description: The distance of sensory deficit to von Frey hairs which measure sensitivity to pressure in centimeters along the transverse horizontal line passing through the anterior superior iliac spine. The von Frey hairs are pushed into the skin along the line described above and moved anterior and posterior until the sensory deficit to pressure is revealed and subsequently measured.
Time Frame: Hourly from Hours 0-6 following the initiation of local anesthetic administration
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Bolus | Basal
Number analyzed (Participants) | 24 | 24
cm
  Hour 0 | 0 (0) | 0 (0)
  Hour 1 | 7.6 (6.0) | 6.0 (8.4)
  Hour 2 | 10.7 (8.3) | 12.2 (9.3)
  Hour 3 | 11.9 (8.2) | 14.5 (5.7)
  Hour 4 | 11.3 (8.6) | 11.6 (7.4)
  Hour 5 | 13.6 (10.0) | 13.4 (7.7)
  Hour 6 | 12.8 (10.0) | 13.2 (7.8)

5. Secondary Outcome: Sensory Deficit (Von Frey Hairs), Mid-axillary Line
Description: The distance of sensory deficit to von Frey hairs which measure sensitivity to pressure in centimeters along the mid-axillary line. The von Frey hairs are pushed into the skin along the line described above and moved cephalad and caudal until the sensory deficit to pressure is revealed and subsequently measured.
Time Frame: Hourly from Hours 0-6 following the initiation of local anesthetic administration
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Bolus | Basal
Number analyzed (Participants) | 24 | 24
cm
  Hour 0 | 0 (0) | 0 (0)
  Hour 1 | 7.4 (6.3) | 3.0 (4.5)
  Hour 2 | 7.4 (4.8) | 6.9 (4.6)
  Hour 3 | 7.9 (6.0) | 9.1 (6.9)
  Hour 4 | 8.8 (7.1) | 7.5 (5.6)
  Hour 5 | 7.8 (6.5) | 10.5 (6.0)
  Hour 6 | 7.0 (5.3) | 6.4 (5.3)

ADVERSE EVENTS:
Time Frame: 7 days
Arm/Group | Bolus | Basal
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 0/24 | 0/24

LIMITATIONS AND CAVEATS:
Lack of surgical pain in the healthy volunteer subjects of this study. Since the subjects of this study were healthy pain-free volunteers, we used cutaneous cold and pressure deficits as surrogate outcome measures.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No